CLINICAL TRIAL: NCT00250770
Title: CSF-1 and Other Cytokines in Human Endometrial Carcinogenesis
Brief Title: Colony-Stimulating Factor-1 (CSF-1) and Other Cytokines in Human Endometrial Carcinogenesis
Status: Withdrawn | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: CSF-1
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Uterine Neoplasms; Endometrial Neoplasms
Keywords: Corpus Uteri; Endometrium; Cancer
MeSH Terms: conditions — Uterine Neoplasms; Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We have collected serum and ascites from approximately 200 patients with endometrial carcinoma and 200 controls. We have long term follow-up serum from approximately 60 of these patients. Approximately 10% of endometrial carcinoma patients recur. Our goal will be to eventually have follow-up serum from up to 60 patients with recurrent endometrial carcinoma in our tissue bank, so that we can determine the role of these assays in predicting recurrence.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Healthy postmenopausal and perimenopausal women with no history of endometrial carcinoma.
  Women undergoing hysterectomy for benign conditions.

SUMMARY:
The purposes of this study are the following:

1. To further characterize and quantify both CSF-1 and colony-stimulating factor-1 receptor (CSF-1R) expression from additional tumor specimens, specifically, tumors of high grade and from metastatic sites.
2. To assay using Enzyme-Linked ImmunoSorbent Assay (ELISA) sandwich monoclonal antibody methodology, CSF-1 expression in the peritoneal fluid and blood from patients with endometrial adenocarcinomas.
3. Using immunohistochemistry, to evaluate the presence of staining for CSF-1 and CSF-1R from additional patients with endometrial adenocarcinomas, especially of high grades and from metastatic sites.
4. To determine the extent of cytokine, specifically CSF-1, but also interleukin-1 (IL-1), IL-6, and granulocyte-macrophage colony-stimulating factor (GM-CSF), production, in endometrial carcinoma cells in primary cell culture.
5. To determine the responsiveness of epithelial cells on estrogen and antiestrogen binding, to determine if CSF-1 production is mediated, in these cells, by estrogen receptor binding, or alternative pathways of intracellular/cell-cell signal transduction.
6. The ultimate objective of these experiments is to characterize CSF-1 expression from benign and tumor cells in order to identify steps in the CSF-1 activated signalling pathways that may represent potential targets for therapy.

DETAILED DESCRIPTION:
These experiments, taken together, should critically determine if there is a role for the CSF-1/ c-fms autocrine, endocrine, or paracrine loop in the progression of endometrial adenocarcinoma. If so, alterations in this loop may provide novel medical therapies for this disease. Additionally, these experiments will determine which are the predominant cytokines expressed in these tumors, and will help the investigators to determine the role, if any, these cytokines play in cancer cell growth and proliferation in relationship with each other and within and outside of the estrogen-mediated pathways.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hysterectomy, or who have endometrial cancer, and are under routine surveillance.
* Patients may have received prior hormonal, cytotoxic chemotherapy, irradiation or surgical therapy.
* Healthy post-menopausal and peri-menopausal women.
* A consent form must be signed by the patient prior to study entry.

Exclusion Criteria:

* Patients who do not have primary uterine corpus tumors.
* Patients with less than one gram of tumor tissue available to procurement.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * All patients undergoing hysterectomy, or who have endometrial cancer, and are under routine surveillance.
  * Patients may have received prior hormonal, cytotoxic chemotherapy, irradiation or surgical therapy.
  * Healthy post-menopausal and peri-menopausal women.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1998-01; Primary Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States